CLINICAL TRIAL: NCT06646523
Title: Effects of Remotely Supervised Home-based High-speed Bodyweight Resistance Training on Bradykinesia in Individuals with Parkinson's Disease: a Randomized Clinical Trial
Brief Title: Effects of Home-based High-speed Bodyweight Resistance Training in Individual with Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Christina Danielli Coelho de Morais Faria, Associate professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 68350023.7.0000.5149
Record Dates: First submitted 2024-10-11; First posted 2024-10-17 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: Exercise; Bradykinesia; Mobility; Rehabilitation; Parkinson disease
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Hypokinesia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-speed bodyweight resistance training (Experimental): The participants of the experimental group (high-speed bodyweight resistance training) will receive a home-based intervention that will include 5 minutes of warm-up (free active movements of trunk and lower limbs), followed by 50 min of exercises more targeted to the lower limb muscles, and by 5 minutes of cool-down (lower limb muscle stretching and relaxation breathing exercise).
  The experimental intervention will be performed at maximum speed. During the initial home visit, the speed at which the participant can perform one set of each exercise at maximum speed will be timed. Speed-based progression will be determined every four weeks by increasing the number of repetitions in each set of exercises performed during subsequent home visits.
  Interventions: Other: High-speed bodyweight resistance training
- Control group (Bodyweight intervention, usual speed) (Sham Comparator): The participants of the control group (Bodyweight intervention, usual speed) will also receive a home-based intervention that will include 5 minutes of warm-up (free active movements of trunk and lower limbs), followed by 50 min of exercises more targeted to the lower limb muscles, and by 5 minutes of cool-down (lower limb muscle stretching and relaxation breathing exercise).
  The control intervention will be performed at the usual speed. The same procedures that will be carried out to determine the maximum speed in the experimental group will be used to determine the usual speed in the control group. There will be no progression in the speed of performing the exercises. However, participants in the control group will also receive a home visit from the main researcher every four weeks to avoid bias related to the amount of attention given to participants in the experimental group.
  Interventions: Other: Control group (Bodyweight intervention, usual speed)

INTERVENTIONS:
Other: High-speed bodyweight resistance training — The participants of the experimental group (high-speed bodyweight resistance training) will receive a home-based intervention that will include 5 minutes of warm-up (free active movements of trunk and lower limbs), followed by 50 min of exercises more targeted to the lower limb muscles, and by 5 minutes of cool-down (lower limb muscle stretching and relaxation breathing exercise).
  The experimental intervention will be performed at maximum speed. During the initial home visit, the speed at which the participant can perform one set of each exercise at maximum speed will be timed. Speed-based progression will be determined every four weeks by increasing the number of repetitions in each set of exercises performed during subsequent home visits.
  Arms: High-speed bodyweight resistance training
Other: Control group (Bodyweight intervention, usual speed) — The participants of the control group (Bodyweight intervention, usual speed) will also receive a home-based intervention that will include 5 minutes of warm-up (free active movements of trunk and lower limbs), followed by 50 min of exercises more targeted to the lower limb muscles, and by 5 minutes of cool-down (lower limb muscle stretching and relaxation breathing exercise).
  The control intervention will be performed at the usual speed. The same procedures that will be carried out to determine the maximum speed in the experimental group will be used to determine the usual speed in the control group. There will be no progression in the speed of performing the exercises. However, participants in the control group will also receive a home visit from the main researcher every four weeks to avoid bias related to the amount of attention given to participants in the experimental group.
  Arms: Control group (Bodyweight intervention, usual speed)

SUMMARY:
Exercises that involve increasing the speed of movements are beneficial for individuals with Parkinson's disease (PD) and have the potential to reduce bradykinesia and improve mobility. High-speed bodyweight resistance training is a treatment that involves increasing speed considered accessible and viable as it can be performed at any time and place, including at home. This treatment has already shown benefits in the elderly individuals, however no studies were found in individuals with PD. Therefore, the primary aim of this study will be to investigate the effects of home-based and remotely supervised high-speed bodyweight resistance training in reducing bradykinesia in individuals with PD. The secondary aim will be to investigate the effects of home-based and remotely supervised high-speed bodyweight resistance training in improving mobility, muscle power, dynamic balance, and quality of life in this population. A randomized controlled trial will be carried out with concealed allocation, blinded assessments, and intention-to-treat analysis. Altogether, 46 individuals with PD (age ≥ 50 years old, who are bradykinetics and sedentary or insufficiently active will be included. Participants will be randomly assigned to either an experimental group (high-speed bodyweight resistance training) or a control group (bodyweight intervention, usual speed). Both groups will perform a home-based and remotely supervised intervention, consisting of 60-min individual sessions, three times per week over 12 weeks, with a trained physiotherapist. Primary outcomes are bradykinesia of the lower limbs and mobility. Secondary outcomes are muscle power, dynamic balance, and quality of life. Between-group differences will be measured by two-way repeated measures ANOVA, considering the baseline, post-training, and 4-week follow-up. The findings of this trial have the potential to provide important insights regarding the effects of high-speed bodyweight resistance training in reducing bradykinesia and improving mobility in individuals with PD. High-speed bodyweight resistance training does not use any type of external resistance and can be performed anywhere and at any time. In addition, it can be performed at home through telemonitoring, reducing time and costs of transport, making it quite feasible and accessible for individuals from different social and economic backgrounds which increases the feasibility of reproducing their findings in clinical practice.

DETAILED DESCRIPTION:
The sample size calculation was performed considering the primary outcome measures bradykinesia (assessed using items 3.8, 3.9, 3.10, and 3.14 of the motor examination of the MDS-UPDRS) based on data provided by previous similar randomized controlled trial. The effect size for bradykinesia was derived from a previous study. In that study, the groups showed a difference in means of -2.3 (treatment effect), using a standard deviation of 2.5, a significance level (α) of 5% and a power of 0.80, a sample size of 40 participants are required. Assuming a dropout rate of 15%, a total of 46 participants will be recruited (23 per group).

All statistical analyses will be performed by an independent examiner, blinded to the group allocation. All data analyses will be performed using SPSS for Windows (SPSS, Chicago, IL, USA). Descriptive statistics will be calculated for all outcomes. The effects of the interventions will be analyzed from the collected data using intention-to-treat. For dropouts, data from the last available assessment will be used for missed sessions. Two-way ANOVA with repeated measures will be used to evaluate the differences between groups, considering the time factor (pre-intervention, post-intervention, and follow-up), followed by post hoc test selected based on final sample size and in the assumption of equal of variance. If necessary, a similar nonparametric test will be used. The level of significance will be set at 5%.

ELIGIBILITY:
Inclusion Criteria

* ≥50 years old;
* Parkinson's disease diagnosed by a neurologista;
* classified between stages 1-3 of the modified Hoehn & Yahr Scale;
* present bradykinesia identified by items 3.8 (Leg Agility) and/or 3.14 (Global Spontaneity of Movement - Body Bradykinesia) of the motor examination of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) with a minimum score of 1 out of 4 points in at least one of the items;
* taking antiparkinsonian medication, and who have been medically stable
* are classified as inactive or insufficiently active; have ability to walk independently without assistive devices; and have written medical permission to allow them to participate in the study. The Centers for Disease Control and Prevention classification will be used to determine if an individual is inactive or insufficiently active. Participants will be asked about the exercises they performed most often over the last 4 weeks, including their frequency and duration. Individuals who report that they have performed physical exercise over the last month at least five times per week for more than 30 min at a moderate intensity or at least three times per week for at least 20 min at a vigorous intensity will be classified as having moderate or vigorous exercise levels, respectively. Individuals who report not having practiced any exercise over the last month will be classified as inactive. Those who report doing physical exercise over the last month that is not classified as vigorous or moderate intensity will be classified as insufficiently active.

Exclusion Criteria:

* cognitive impairments as determined by cutoff scores (in points) of the Mini-Mental Status Examination according to education level reference;
* any other neurological, musculoskeletal, cardiovascular, or respiratory disorders that could affect their ability to perform the tests;
* used deep brain stimulation (DBS);
* no access to the internet;
* who do not have a caregiver or family member who can assist during the intervention sessions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Bradykinesia - Unified Parkinson's Disease Rating Scale | At baseline, 12 weeks post-intervention, and at 4-week follow-up
  Bradykinesia will be measured by items 3.8 (Leg Agility), 3.9 (Arising From Chair), 3.10 (Gait), and 3.14 (Global Spontaneity of Movement - Body Bradykinesia) of the motor examination of the Unified Parkinson's Disease Rating Scale. Each item is scored '0'- '4' on a categorical scale, with '0' indicating the absence of the symptom or normal activity and '4' indicating the presence of the symptom or deficit. Higher scores indicate severe bradykinesia

SECONDARY OUTCOMES:
Change from baseline in Mobility - 10-m walk test | At baseline, 12 weeks post-intervention, and at 4-week follow-up
  Mobility will be measured using the 10-m walk test. Participants will be instructed to walk at both comfortable and maximal speeds in a 14-m hallway and the time taken to cover the central 10-m will be timed. A digital stopwatch will be used to measure three comfortable and maximal speeds measurements. The average of the three measurements will be used for analysis.
Change from baseline in Muscle power - Five Time Sit to Stand | At baseline, 12 weeks post-intervention, and at 4-week follow-up
  Muscle power will be assessed using Five Time Sit to Stand. Participants will be instructed to perform five time sit to stand repetitions as rapidly as possible using a chair without armrests and with a standardized height. The time needed to complete the task will be recorded with a stopwatch. Only one repetition will be performed after one or two familiarization. Mean muscle power will be obtained by the product of mean velocity and mean force.
Change from baseline in Dynamic balance - Mini-Balance Evaluation System's Test | At baseline, 12 weeks post-intervention, and at 4-week follow-up
  Dynamic balance will be assessed using Mini-Balance Evaluation System's Test. This test assesses changes in balance representing four domains of dynamic balance: anticipatory postural adjustments, postural responses, sensory orientation, and dynamic gait. The Mini-Balance Evaluation System's Test is composed of 14 items, and for each item, the scores range from 0 to 2. A higher score indicates better performance.
Change from baseline in Quality of life - Parkinson's Disease Questionnaire-39 | At baseline, 12 weeks post-intervention, and at 4-week follow-up
  Quality of life will be measured using Parkinson's Disease Questionnaire-39. The Parkinson's Disease Questionnaire-39 is composed of 39 items divided into eight dimensions: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. The score for each item ranges from 0 to 4, and for each dimension varies from 0 to 100. A higher score indicates worse the individual's perception of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Christina CM Faria, Ph.D., Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing. 1997 Sep;26(5):353-7. doi: 10.1093/ageing/26.5.353. PMID 9351479
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Background] Alcazar J, Losa-Reyna J, Rodriguez-Lopez C, Alfaro-Acha A, Rodriguez-Manas L, Ara I, Garcia-Garcia FJ, Alegre LM. The sit-to-stand muscle power test: An easy, inexpensive and portable procedure to assess muscle power in older people. Exp Gerontol. 2018 Oct 2;112:38-43. doi: 10.1016/j.exger.2018.08.006. Epub 2018 Sep 1. PMID 30179662
- [Background] Lim LI, van Wegen EE, de Goede CJ, Jones D, Rochester L, Hetherington V, Nieuwboer A, Willems AM, Kwakkel G. Measuring gait and gait-related activities in Parkinson's patients own home environment: a reliability, responsiveness and feasibility study. Parkinsonism Relat Disord. 2005 Jan;11(1):19-24. doi: 10.1016/j.parkreldis.2004.06.003. PMID 15619458
- [Background] Bertolucci PH, Brucki SM, Campacci SR, Juliano Y. [The Mini-Mental State Examination in a general population: impact of educational status]. Arq Neuropsiquiatr. 1994 Mar;52(1):1-7. Portuguese. PMID 8002795
- [Background] Centers for Disease Control and Prevention (CDC). Physical activity trends--United States, 1990-1998. MMWR Morb Mortal Wkly Rep. 2001 Mar 9;50(9):166-9. PMID 11393487
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Vasconcellos LS, Silva RS, Pacheco TB, Nagem DA, Sousa CO, Ribeiro TS. Telerehabilitation-based trunk exercise training for motor symptoms of individuals with Parkinson's disease: A randomized controlled clinical trial. J Telemed Telecare. 2023 Oct;29(9):698-706. doi: 10.1177/1357633X211021740. Epub 2021 Jun 18. PMID 34142896
- [Background] Lai B, Rimmer J, Barstow B, Jovanov E, Bickel CS. Teleexercise for Persons With Spinal Cord Injury: A Mixed-Methods Feasibility Case Series. JMIR Rehabil Assist Technol. 2016 Jul 14;3(2):e8. doi: 10.2196/rehab.5524. PMID 28582252
- [Background] Jaque C, Veliz P, Ramirez-Campillo R, Moran J, Gentil P, Cancino J. High-Speed Bodyweight Resistance Training Improves Functional Performance Through Maximal Velocity in Older Females. J Aging Phys Act. 2021 Aug 1;29(4):659-669. doi: 10.1123/japa.2020-0129. Epub 2020 Dec 25. PMID 33361494
- [Background] Jaque-Gallardo C, Veliz-Campillay P, Cancino-Lopez J. [Effect of a high-speed bodyweight resistance training on timed up and go and one leg stance in older women]. Rev Med Chil. 2019 Sep;147(9):1136-1143. doi: 10.4067/s0034-98872019000901136. Spanish. PMID 33625447
- [Background] Ni M, Signorile JF, Mooney K, Balachandran A, Potiaumpai M, Luca C, Moore JG, Kuenze CM, Eltoukhy M, Perry AC. Comparative Effect of Power Training and High-Speed Yoga on Motor Function in Older Patients With Parkinson Disease. Arch Phys Med Rehabil. 2016 Mar;97(3):345-354.e15. doi: 10.1016/j.apmr.2015.10.095. Epub 2015 Nov 4. PMID 26546987
- [Background] Ni M, Signorile JF, Balachandran A, Potiaumpai M. Power training induced change in bradykinesia and muscle power in Parkinson's disease. Parkinsonism Relat Disord. 2016 Feb;23:37-44. doi: 10.1016/j.parkreldis.2015.11.028. Epub 2015 Nov 27. PMID 26698015
- [Background] Ridgel AL, Ault DL. High-Cadence Cycling Promotes Sustained Improvement in Bradykinesia, Rigidity, and Mobility in Individuals with Mild-Moderate Parkinson's Disease. Parkinsons Dis. 2019 Mar 3;2019:4076862. doi: 10.1155/2019/4076862. eCollection 2019. PMID 30944720
- [Background] Uygur M, Bellumori M, LeNoir K, Poole K, Pretzer-Aboff I, Knight CA. Immediate effects of high-speed cycling intervals on bradykinesia in Parkinson's disease. Physiother Theory Pract. 2015 Feb;31(2):77-82. doi: 10.3109/09593985.2014.972530. Epub 2014 Oct 27. PMID 25347790
- [Background] Bologna M, Paparella G, Fasano A, Hallett M, Berardelli A. Evolving concepts on bradykinesia. Brain. 2020 Mar 1;143(3):727-750. doi: 10.1093/brain/awz344. PMID 31834375
- [Background] Morris ME. Movement disorders in people with Parkinson disease: a model for physical therapy. Phys Ther. 2000 Jun;80(6):578-97. PMID 10842411
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468